CLINICAL TRIAL: NCT00829660
Title: A Long-term, Multicentre, Double-blind, Randomised Parallel-group Trial to Determine Whether Reducing Post-prandial Glycaemia Can Reduce Cardiovascular-related Morbidity and Mortality in Patients With Established Coronary Heart Disease or Acute Coronary Syndrome Who Have Impaired Glucose Tolerance
Brief Title: Acarbose Cardiovascular Evaluation Trial
Acronym: ACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11232; ISRCTN91899513
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Coronary Heart Disease; Acute Coronary Syndrome; Impaired Glucose Tolerance; Type 2 Diabetes Mellitus (T2DM)
Keywords: Acarbose
MeSH Terms: conditions — Coronary Disease; Acute Coronary Syndrome; Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Acarbose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acarbose (Active Comparator): The participants were given one tablet (50mg) of acarbose per day, taken with a meal during their first week (7 days). During the second week, the dose was increased to two tablets/day (50mg twice a day i.e. 100mg/day) and then three tablets/day (50mg three times a day i.e. 150mg/day) thereafter. The maximum tolerated dose is being taken for the duration of the trial (maximum dose is 150mg/day).
  Interventions: Drug: Acarbose
- Matching Placebo (Placebo Comparator): The participants were given one tablet of matching placebo per day, taken with a meal during their first week (7 days). During the second week, the dose was increased to two tablets/day and then three tablets/day thereafter. The maximum tolerated dose is being taken for the duration of the trial (maximum dose is 3 tablets/day).
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Acarbose — The participants were given one tablet (50mg) of acarbose per day, taken with a meal during their first week (7 days). During the second week, the dose was increased to two tablets/day (50mg twice a day i.e. 100mg/day) and then three tablets/day (50mg three times a day i.e. 150mg/day) thereafter. The maximum tolerated dose is being taken for the duration of the trial (maximum dose is 150mg/day).
  Other Names: Glucobay
  Arms: Acarbose
Drug: Matching Placebo — The participants were given one tablet of matching placebo per day, taken with a meal during their first week (7 days). During the second week, the dose was increased to two tablets/day and then three tablets/day thereafter. The maximum tolerated dose is being taken for the duration of the trial (maximum dose is 3 tablets/day).
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to determine whether acarbose therapy can reduce cardiovascular-related morbidity and mortality in patients with impaired glucose tolerance (IGT) who have established coronary heart disease (CHD) or acute coronary syndrome (ACS). A secondary objective of the study is to determine if acarbose therapy can prevent or delay transition to type 2 diabetes mellitus (T2DM) in this patient population.

DETAILED DESCRIPTION:
A long-term, multicentre, double-blind, randomised parallel-group trial to determine whether reducing post-prandial glycaemia can reduce cardiovascular-related morbidity and mortality in patients with established coronary heart disease or acute coronary syndrome who have impaired glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 50 years or more.
* Definite CHD, defined as a, b or c below:

  1. Previous myocardial infarction (MI) or Acute Coronary Syndrome (ACS), but not within the last 3 months, with any two of the following:

     * Typical clinical presentation
     * Confirmatory ECG changes
     * Appropriate elevation of cardiac enzymes/biomarkers
  2. Previous unstable angina (UA) or Acute Coronary Syndrome (ACS), but not within the last 3 months, with any two of the following:

     * Typical clinical presentation
     * Confirmatory ECG changes
     * Either elevation of a cardiac biomarker or a >50% stenosis in ≥1 major epicardial coronary artery shown on coronary angiography or CT angiography. Where stenosis is reported in a qualitative manner, the categories "moderate" and "severe" will be taken as equating to >50% stenosis.
  3. Current stable angina defined as:

     * Typical clinical history with symptoms occurring within the last month, and
     * A >50% stenosis in ≥1 major epicardial coronary artery shown on coronary angiography or CT angiography. Where stenosis is reported in a qualitative manner, the categories "moderate" and "severe" will be taken as equating to >50% stenosis.
* Impaired glucose tolerance diagnosed on a single standard oral glucose tolerance test (OGTT) , defined as a 2-hour plasma glucose (2HPG) value ≥7.8 but <11.1 mmol/l and a fasting plasma glucose (FPG) <7.0 mmol/l within six months prior to enrollment.
* Optimised cardiovascular drug therapy.
* At least 80% adherent to single blind placebo Study Medication during the run-in period.
* Provision of written informed consent.

Exclusion Criteria:

* Previous history of diabetes, other than gestational diabetes.
* MI, unstable angina, stroke or a transient ischaemic attack (TIA) within the previous three months.
* Planned or anticipated coronary, cerebrovascular or peripheral arterial revascularisation or other major surgical intervention, at the time of randomisation
* New York Heart Association (NYHA) class III or IV heart failure.
* Evidence of severe hepatic disease.
* Evidence of severe renal impairment or an eGFR <30 ml/min/1.73m2 (derived using the Modification of Diet in Renal Disease, MDRD, Chinese equation)
* Any other condition likely to reduce adherence to the protocol e.g. alcoholism, major active psychiatric disorder, cognitive impairment or a condition likely to markedly limit life expectancy e.g. malignancy.
* Pregnancy (or planned pregnancy within the next five years).
* Concurrent participation in any other clinical interventional trial. Note: Patients who were treated previously with an alphaglucosidase inhibitor must have at least a three-month washout period before being randomised into the ACE trial.
* Known intolerance to alpha glucosidase inhibitors or gastrointestinal problems.
* Thought by the investigator for any reason to be unsuitable for participation in this clinical study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6526 (Actual)
Dates: Start 2009-02-17 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
A composite cardiovascular outcome defined as the time after randomisation to the first occurrence of any one of the following: -Cardiovascular death -Non-fatal MI -Non-fatal stroke -Hospitalisation for Unstable Angina -Hospitalisation for Heart Failure | Follow-up until 728 adjudicated Primary Outcome Measures have been recorded

SECONDARY OUTCOMES:
Transition to type 2 diabetes confirmed by two successive diagnostic plasma glucose values (FPG >7.0 mmol/l and/or 2HPG > 11.1 mmol/l), with no intervening non-diagnostic values.
All cause mortality
Each of the components of the primary composite cardiovascular outcome will also be analysed individually, both as first and as total events.
Major Cardiovascular Event (MACE) composite cardiovascular outcome, defined as the time after randomisation to the first occurrence of any one of the following: - Cardiovascular death - Non-fatal MI - Non-fatal stroke
Impaired renal function as evidenced by: A reduced estimate of glomerular filtration rate( eGFR <30 ml/minute/ 1.73 m2) estimated using the Chinese MDRD formula, a doubling of the baseline plasma creatinine level, a halving of the baseline eGFR
Resource use, costs and cost effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Professor Rury R Holman, FRCP FMedSci, Principal Investigator — Diabetes Trials Unit, University of Oxford
Locations (176):
- China (175):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chuiyangliu Hospital, Beijing, Beijing Municipality
  - China Meitan General Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital of The Capital University of Medical Sciences, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Ji Shui Tan Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Fu Xing Hospital, Beijing, Beijing Municipality
  - Beijing Shijingshan Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Aerospace Central Hospital, Beijing, Beijing Municipality
  - Affiliated to The Capital University of Medical Sciences Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Wangjing Hospital of CACMS, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Healthy Palace Hospital, Beijing, Beijing Municipality
  - Aerospace 731 Hospital, Beijing, Beijing Municipality
  - General Hospital of Second Artillery PLA, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - PLA General Hospital, Beijing, Beijing Municipality
  - Anzhen Hospital of The Capital University of Medical Sciences 2nd., Beijing, Beijing Municipality
  - Beijing Pinggu Hospital, Beijing, Beijing Municipality
  - Beijing Yanhua Hospital, Beijing, Beijing Municipality
  - Chongqing Medical University Second Afflicated Hospital, Chongqing, Chongqing Municipality
  - Chongqing Zhongshan Hospital, Chongqing, Chongqing Municipality
  - Chongqing Third People's Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Da Ping Hospital, Chongqing, Chongqing Municipality
  - The Second People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Union Hospital Affiliated to Fujian Medical University, Fuzhou, Fujian
  - The People's Hospital of Fujian Province, Fuzhou, Fujian
  - The First Hospital of Xiamen, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Wu Jing Zhong Dui Hospital of Guangdong Province, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Zhong Shan City People's Hospital, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-Sen University, Zhuhai, Guangdong
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Minzu Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - 303 Hospital of People's Liberation Army, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Bethune International Peace Hospital, Shijiazhuang, Hebei
  - Tangshan Workers Hospital, Tangshan, Hebei
  - The Affiliated Hospital of North China Coal Medical University, Tangshan, Hebei
  - Yu Tian County Hospital, Tangshan, Hebei
  - The Third Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - Da Qing Oilfield General Hospital, Daqing, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan Science & Technology University, Luoyang, Henan
  - Luo Yang Central Hospital, Affiliated to Zhengzhou University, Luoyang, Henan
  - The First Affiliated Hospital of Henan College of TCM, Zhengzhou, Henan
  - The People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College of Huazhong, Wuhan, Hubei
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College of Huazhong, Wuhan, Hubei
  - Pu'ai Hospital of Wuhan City, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Fourth Hospital of Changsha, Changsha, Hunan
  - Xiangya Hospital Central-South University, Changsha, Hunan
  - The Third Hospital of Changsha, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - Inner Mongolia Hospital, Hohhot, Inner Mongolia
  - 81st Hospital of Chinese PLA, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Nanjing Zhongda Hospital, Nanjing, Jiangsu
  - BENQ Hospital, Nanjing, Jiangsu
  - Jiangsu Province Official Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jiangsu Provincial Hospital of TCM, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Wuxi No.3 People's Hospital, Wuxi, Jiangsu
  - Hospital Affiliated Xuzhou Medical University, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Zhenjiang First People's Hospital, Zhenjiang, Jiangsu
  - Jiujiang University Hospital, Jiujiang, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Third Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The Central Hospital of Anshan, Anshan, Liaoning
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - The First Hospital of Dalian Medical University, Dalian, Liaoning
  - Dalian Central Hospital, Dalian, Liaoning
  - Xianyang Central Hospital, Shengyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - The Fourth Hospital of China Medical University, Shenyang, Liaoning
  - The First Hospital of Yinchuan, Yinchuan, Ningxia
  - Affiliated Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Xi'an Central Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Affiliated Hospital of Xi'an Medical college, Xi'an, Shaanxi
  - Affiliated Hospital of Yan'an University, Yan’an, Shaanxi
  - Yan'an People's Hospital, Yan’an, Shaanxi
  - The First Hospital of Yulin, Yulin, Shaanxi
  - The Central Hospital of Jinan, Jinan, Shandong
  - The First People's Hospital of Jinan, Jinan, Shandong
  - The General Hospital of Jinan Military Region, Jinan, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Hospital Affiliated of Medical School, Qingdao University, Qingdao, Shandong
  - The Qingdao Municiple Hospital, Qingdao, Shandong
  - Qingdao Fuwai Hospital, Shibei, Shandong
  - Taian City Central Hospital, Taian, Shandong
  - Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital Affiliated to the Shanghai Jiaotong University Medical School, Shanghai, Shanghai Municipality
  - Shanghai Central Hospital of Xuhui District, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Huadong Hospital, Shanghai, Shanghai Municipality
  - Shanghai Putuo District People's Hospital, Shanghai, Shanghai Municipality
  - Putuo District Center Hospital, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Number 411 Hospital of PLA, Shanghai, Shanghai Municipality
  - Shanghai Central Hospital of Yangpu District, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital Affilicated to Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area Gongli Hospital, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai Zhabei District Shibei Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jinshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong New District People's Hospital, Shanghai, Shanghai Municipality
  - General Hospital of Tisco, Taiyuan, Shanxi
  - The Third Engineering Bureau Hospital of Ministry of Railway, Taiyuan, Shanxi
  - Taiyuan City Central Hospital, Taiyuan, Shanxi
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - PLA No.323 Hospital, Xi’an, Shanxi
  - Chengdu First People's Hospital, Chengdu, Sichuan
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The West China Hospital, Chengdu, Sichuan
  - Sichuan Mianyang 404 Hospital, Sichuan, Sichuan
  - Tianjin Union Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin Union Medicine Centre, Tianjin, Tianjin Municipality
  - Army Police's Medical College Affiliated Hospital, Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Center Hospital, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Dagang Oil-Field General Hospital, Tianjin, Tianjin Municipality
  - The Fifth Central Hospital of Tianjin, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of the Medical College, Shihezi, Xinjiang
  - Xin Jiang Traditional Chinese Medicine Hospital, Ürümqi, Xinjiang
  - General Hospital of Xinjiang Production and Construction Corps, Ürümqi, Xinjiang
  - The 474th Hospital of PLA, Ürümqi, Xinjiang
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical College, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Second Affiliated Hospital of Kunming Medical College, Kunming, Yunnan
  - People's Hospital of Yuxi City, Yuxi, Yunnan
  - Zhe Jiang Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Affiliated With School of Medicine, Zhe Jiang University, Hangzhou, Zhejiang
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wamil M, McMurray JJV, Scott CAB, Coleman RL, Sun Y, Standl E, Ryden L, Holman RR. Predicting heart failure events in patients with coronary heart disease and impaired glucose tolerance: Insights from the Acarbose Cardiovascular Evaluation (ACE) trial. Diabetes Res Clin Pract. 2020 Dec;170:108488. doi: 10.1016/j.diabres.2020.108488. Epub 2020 Oct 6. PMID 33035598
- [Derived] Gerstein HC, Coleman RL, Scott CAB, Xu S, Tuomilehto J, Ryden L, Holman RR; ACE Study Group. Impact of Acarbose on Incident Diabetes and Regression to Normoglycemia in People With Coronary Heart Disease and Impaired Glucose Tolerance: Insights From the ACE Trial. Diabetes Care. 2020 Sep;43(9):2242-2247. doi: 10.2337/dc19-2046. Epub 2020 Jul 8. PMID 32641379
- [Derived] Holman RR, Coleman RL, Chan JCN, Chiasson JL, Feng H, Ge J, Gerstein HC, Gray R, Huo Y, Lang Z, McMurray JJ, Ryden L, Schroder S, Sun Y, Theodorakis MJ, Tendera M, Tucker L, Tuomilehto J, Wei Y, Yang W, Wang D, Hu D, Pan C; ACE Study Group. Effects of acarbose on cardiovascular and diabetes outcomes in patients with coronary heart disease and impaired glucose tolerance (ACE): a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2017 Nov;5(11):877-886. doi: 10.1016/S2213-8587(17)30309-1. Epub 2017 Sep 13. PMID 28917545
- See also: Diabetes Trials Unit, International Co-ordinating Centre for the ACE Trial — http://www.dtu.ox.ac.uk/ACE